CLINICAL TRIAL: NCT03860142
Title: Evolution of Food Orality in Children Aged Between 24 and 36 Months: Comparison of the Severity and Specificities of Disorders Between Two Populations of Children, Born Very Prematurely and Born at Term
Acronym: EvOral
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 18-PP-06
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Infant, Premature, Diseases
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- full-term child born: use of a new scale to rate the severity of food disorders on full-term child born
  Interventions: Behavioral: Archet scale
- premature child born: use of a new scale to rate the severity of food disorders on premature child born
  Interventions: Behavioral: Archet scale

INTERVENTIONS:
Behavioral: Archet scale — Parents will be asked to answer questions about their child's nutrition by using a new scale : Archet scale

SUMMARY:
Oral disorders are currently widely described in the premature birth population, but few studies compare them to their prevalence in the full-term population.

In addition, new behaviours and eating habits are regularly emerging in our society.

The objective of this study is to compare the severity of signs of oral disorders between the group of preterm infants and the group of term infants born without organic pathologies that compromise oral development.

ELIGIBILITY:
Inclusion Criteria:

* Children whose age ≥ 24 months and ≤ 36 months
* Full-term or prematurely born (<33 SA) at Nice University Hospital

Exclusion Criteria:

* Children with congenital pathologies (with malformations in the oro-facial sphere)
* Children with neurological and developmental pathologies unrelated to prematurity
* Children with ENT deformities
* Parental langage barrier

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: term and prematurely born child
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Archet scale score | 15 mn
  The severity of the signs of food orality disorders is assessed by Archet Scale, which makes it possible to establish a score out of 20. The severity of the signs is divided into four classes according to the following scores: from 0 to 5 = zero to low grade, from 6 to 10 = light grade, from 11 to 15 = moderate grade, from 16 to 20 = severe grade

CONTACTS AND LOCATIONS:
Locations (1):
- Nice hospital, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided